CLINICAL TRIAL: NCT03988166
Title: Chronic Total Occlusion Percutaneous Coronary Intervention CTO-PCI Study
Brief Title: Chronic Total Occlusion Percutaneous Coronary Intervention Study
Acronym: CTO-PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Solutions LLC (Industry)
Collaborators: Teleflex (Industry); Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST2955
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2021-10

CONDITIONS: Chronic Total Occlusion; Ischemic Heart Disease; Chronic Total Occlusion of Coronary Artery
Keywords: Chronic Total Occlusion; Percutaneous revascularization
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, single-arm, intent-to-treat, literature-controlled clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Chronic Total Occlusion Percutaneous Coronary Intervention (Other): CTO percutaneous coronary intervention (PCI) in which at least one Teleflex guidewire and at least one Turnpike catheter are used.
  Interventions: Procedure: Chronic Total Occlusion Revascularization; Device: GuideLiner® V3 catheter, TrapLiner® catheter, Turnpike® catheter

INTERVENTIONS:
Procedure: Chronic Total Occlusion Revascularization — Teleflex's series of study guidewires and catheters will be used to facilitate the safe and effective crossing of de novo CTOs and placement of conventional guidewires beyond the lesion via either a true lumen or subintimal pathway.
Device: GuideLiner® V3 catheter, TrapLiner® catheter, Turnpike® catheter — GuideLiner® V3 catheter, TrapLiner® catheter, Turnpike® catheter

SUMMARY:
The objective of this study is to evaluate angiographic confirmation of placement of any guidewire beyond the CTO, in the true vessel lumen, in patients undergoing CTO percutaneous coronary intervention (PCI) in which at least one Teleflex guidewire and at least one Turnpike catheter are used.

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm, intent-to-treat, literature-controlled clinical study. The study will be conducted in up to 15 investigational sites in the U.S. This study will enroll up to 150 patients to provide adequate powering for hypothesis testing and an evaluable sample size of at least 135 patients.

The population for this study is participants with signs and/or symptoms considered typical of ischemic heart disease attributed to a de novo CTO in a native coronary artery who are suitable candidates for a percutaneous revascularization.

Study devices include the GuideLiner® V3 catheter, TrapLiner® catheter, Turnpike® catheter, and a series of five coronary guidewires (SpectreTM guidewire, R350TM guidewire, RaiderTM guidewire, WarriorTM guidewire, and BanditTM guidewire). All study devices are currently 510(k) cleared for non-CTO indications.

* GuideLiner catheters are intended to be used in conjunction with guide catheters to access discrete regions of the coronary and/or peripheral vasculature, to facilitate placement of interventional devices, and to assist in crossing de novo chronic total occlusions (CTO).
* The TrapLiner catheter is intended for use in conjunction with guide catheters to access discrete regions of the coronary and/or peripheral vasculature, to facilitate placement of interventional devices, to facilitate the exchange of an interventional device while maintaining the position of a guidewire within the vasculature, and to assist in crossing de novo chronic total occlusions (CTO).
* The Turnpike catheters are intended to be used to access discrete regions of the coronary and/or peripheral vasculature. They may be used to facilitate placement and exchange of guidewires, to subselectively infuse/deliver diagnostic and therapeutic agents, and to assist in crossing de novo coronary chronic total occlusions (CTO). The Teleflex guidewires are intended for use in percutaneous procedures to introduce and position catheters and other interventional devices within the coronary and peripheral vasculature, including use in crossing or assisting in crossing de novo coronary chronic total occlusions (CTO).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria:

General inclusion criteria

1. At least 18 years of age at the time of consent
2. Experiencing clinical symptoms considered suggestive of ischemic heart disease (e.g., chest pain or discomfort, heart failure) or has evidence of myocardial ischemia (e.g., abnormal functional study) attributed to the CTO target vessel and is scheduled for clinically indicated percutaneous revascularization
3. Participant is eligible and consents to undergo PCI procedure
4. Acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergency coronary artery bypass grafting (CABG)
5. Willing and able to sign a study Informed Consent Form (ICF) approved by a local or central Institutional Review Board (IRB)
6. Female participants of childbearing potential must have a negative pregnancy test per standard of care for PCI and be practicing contraception

   Angiographic inclusion criteria
7. A minimum of one de novo lesion with at least one target segment in a native coronary vessel meeting the definition of CTO (any non-acute total coronary occlusion fulfilling the angiographic characteristics consistent with high-grade native coronary stenosis (Thrombolysis in Myocardial Infarction (TIMI) score of 0 or 1) and estimated to be in duration of ≥ 3 months by clinical history and/or comparison with antecedent angiogram or electrocardiogram)

Exclusion Criteria:

Participants must not meet any of the following exclusion criteria:

General exclusion criteria

1. History of allergy to iodinated contrast that cannot be effectively managed medically
2. Evidence of acute myocardial infarction (MI) within 72 hours prior to the intended treatment defined as creatine kinase-muscle brain subunits (CK-MB) greater than 3 times the upper limit of normal (ULN)
3. Previous coronary interventional procedure of any kind within 30 days prior to the procedure
4. Any contraindication to cardiac catheterization or to any of the standard concomitant therapies used during routine cardiac catheterization and PCI (e.g., aspirin, clopidogrel, unfractionated heparin)
5. Target lesion requires treatment with another device, after successful crossing with a study device, other than PTCA devices prior to stent placement
6. Atherectomy procedure is planned for the target lesion
7. Known history of clinically significant abnormal laboratory findings ≤ 14 days prior to enrollment, including:

   * Neutropenia (<1000 neutrophils/mm^3)
   * Thrombocytopenia (<100,000 platelets/mm^3)
   * Aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase, or bilirubin > 1.5 × ULN
   * Serum creatinine >2.0 mg/dL
8. Evidence of current clinical instability including the following:

   * Sustained systolic blood pressure <100 mmHg or cardiogenic shock
   * Acute pulmonary edema or severe congestive heart failure (CHF). Severe CHF is defined as New York Heart Association (NYHA) Class IV
   * Suspected acute myocarditis, pericarditis, endocarditis, or cardiac tamponade
   * Suspected dissecting aortic aneurysm
   * Hemodynamically significant valvular heart disease, hypertrophic cardiomyopathy, restrictive cardiomyopathy, or congenital heart disease
9. History of stroke or transient ischemic attack within 6 months prior to procedure
10. Active peptic ulcer or upper gastrointestinal bleeding within 6 months prior to procedure
11. History of bleeding diathesis or coagulopathy or refusal of blood transfusions
12. Other pathology such as cancer, known mental illness, etc., which might, in the opinion of the Investigator, put the patient at risk or confound the results of the study
13. Unable or unwilling to comply with the protocol
14. Currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; or requires coronary angiography, intravascular ultrasound, or other coronary artery imaging procedures

    Angiographic exclusion criteria
15. Occlusion involves segment within previous stent ("in-stent occlusions")
16. Extensive lesion-related thrombus (TIMI thrombus grade 3 or 4)
17. Previous stenting (drug-eluting or bare metal) in the target vessel unless the following conditions are met:

    * It has been at least 9 months since the previous stenting
    * Target lesion is ≥15 mm away from the previously placed stent
    * Previously stented segment (stent plus 5 mm on either side) has no more than 40 percent diameter stenosis, based on visual estimate
18. Target vessel has other lesions proximal to the total occlusion identified with > 75 percent diameter stenosis based on visual estimate; exception: planned stenting of a lesion proximal to the target lesion that can be covered by a single stent (i.e., tandem lesions) is acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Kandzari, MD, Principal Investigator — Piedmont Heart Institute; Dimitrios Karmpaliotis, MD, PhD, Principal Investigator — Columbia University
Locations (13):
- United States (13):
  - Torrance Memorial Medical Center, Torrance, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kandzari DE, Alaswad K, Jaffer FA, Brilakis E, Croce K, Kearney K, Spaedy A, Yeh R, Thompson C, Nicholson W, Wyman RM, Riley R, Lansky A, Buller C, Karmpaliotis D. Safety and efficacy of dedicated guidewire, microcatheter, and guide catheter extension technologies for chronic total coronary occlusion revascularization: Primary results of the Teleflex Chronic Total Occlusion Study. Catheter Cardiovasc Interv. 2022 Feb;99(2):263-270. doi: 10.1002/ccd.29962. Epub 2021 Sep 28. PMID 34582080

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Total Occlusion Percutaneous Coronary Intervention
Started | 150
Completed | 147
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Evaluation of procedural and in-hospital outcomes among 150 patients undergoing attempted CTO revascularization utilizing specialized guidewires, microcatheters and guide extensions.
Arm/Group | Chronic Total Occlusion Percutaneous Coronary Intervention
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 8
  White | 130
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedure Success
Description: Defined as angiographic visualization of any guidewire in a position either distal or proximal to the occlusion depending on the route of access and the absence of in-hospital major adverse cardiac events (MACE).
  • MACE defined as any serious adverse experience that includes cardiac death, target lesion revascularization, or post-procedural myocardial infarction (MI) (Q-wave or non-Q-wave, with creatine kinase (CK) with Muscle (M)-Brain (B) subunits > 3 ULN).
Time Frame: Through Discharge up to 24 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Total Occlusion Percutaneous Coronary Intervention
Number analyzed (Participants) | 150
Participants | 121

2. Secondary Outcome: Number of Participants With Successful Recanalization.
Description: Defined as angiographic confirmation of crossing the chronic total occlusion and restoring blood flow to the affected area.
Time Frame: Through Procedure, up to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Total Occlusion Percutaneous Coronary Intervention
Number analyzed (Participants) | 150
Participants | 142

3. Secondary Outcome: Number of Participants With In-hospital MACE.
Description: Defined as any serious adverse experience that includes cardiac death, target lesion revascularization, or post-procedural MI (Q-wave or non-Q-wave, with CK-MB > 3 ULN). The components of MACE will also be reported separately.
Time Frame: Through Discharge up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Total Occlusion Percutaneous Coronary Intervention
Number analyzed (Participants) | 150
Participants | 29

4. Secondary Outcome: Number of Participants With Clinically Significant Perforation.
Description: Defined as any perforation resulting in hemodynamic instability and/or requiring intervention including pericardiocentesis, embolization, prolonged balloon occlusion, stent graft, or comparable therapy.
Time Frame: Through Procedure up to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Total Occlusion Percutaneous Coronary Intervention
Number analyzed (Participants) | 150
Participants | 16

5. Secondary Outcome: Number of Participants With Procedural Success According to Crossing Technique.
Description: Procedural success is defined as angiographic visualization of any guidewire in a position either distal or proximal to the occlusion depending on the route of access and the absence of in-hospital major adverse cardiac events (MACE).
Time Frame: Through Procedure up to 4 hours post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- Antegrade: CTO percutaneous coronary intervention (PCI) in which at least one Teleflex guidewire and at least one Turnpike catheter are used using the Antegrade approach/technique.
- Retrograde: CTO percutaneous coronary intervention (PCI) in which at least one Teleflex guidewire and at least one Turnpike catheter are used using the retrograde approach/technique.
- Combined Antegrade and Retrograde: CTO percutaneous coronary intervention (PCI) in which at least one Teleflex guidewire and at least one Turnpike catheter are used using both antegrade and retrograde approaches/techniques.
Arm/Group | Antegrade | Retrograde | Combined Antegrade and Retrograde
Number analyzed (Participants) | 81 | 2 | 67
Participants | 69 | 1 | 43

6. Secondary Outcome: Number of Participants With Technical Success.
Description: Defined as successful guidewire recanalization is applicable to investigational devices as at least one investigational guidewire must be used in every procedure.
Time Frame: Through Procedure up to 4 hours post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Total Occlusion Percutaneous Coronary Intervention
Number analyzed (Participants) | 150
Participants | 140

ADVERSE EVENTS:
Time Frame: Collection of Adverse Events (AE) occurred after enrollment through end of the study participation (30-days)
Arm/Group | Chronic Total Occlusion Percutaneous Coronary Intervention
All-Cause Mortality (participants affected / at risk) | 1/150
Serious Adverse Events (participants affected / at risk) | 38/150
Other Adverse Events (participants affected / at risk) | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Total Occlusion Percutaneous Coronary Intervention (N=150)
Myocardial Infarction (MI) (Cardiac disorders) | 27 (27) — CK MB ≥ three times (3X) ULN
Myocardial Infarction (Cardiac disorders) | 9 (9) — CK MB ≥ ten times (10X) ULN
Death (Cardiac disorders) | 1 (1) — Cardiac Death
Target Lesion Revascularization (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT03988166/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT03988166/SAP_001.pdf